CLINICAL TRIAL: NCT00584792
Title: Diet, Genetic Variation and Prostate Cancer Among African Americans
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Lesley Butler, PhD, University of California, Davis
Other Study IDs: 200614379; AA Pilot Study
Record Dates: First submitted 2007-12-22; First posted 2008-01-02 (Estimated); Last update posted 2008-01-02 (Estimated); Status verified 2007-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum collected for Ancestry Imformative Markers (AIMS) testing along with PSA and CRP.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Controls (No prostate cancer)
- 2: Cases (Prostate Cancer Diagnosed)

SUMMARY:
This is a single center pilot study to asses the feasibility of conducting a larger population-based study. It is an investigator-initiated study funded yb the UC Davis Cancer Center's Development Award Program. The hypothesis is that the percent african ancestry in an individual may determine their prognosis if diagnosed with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

Self-identification as a male with African ancestry Between ages of 35-75

Exclusion Criteria:

No African ancestry Not between ages of 35-75

-

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African American males between the ages of 35 and 75.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2006-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Is there a difference in ancestry percentage between the controls (no cancer) and the cases (prostate cancer) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Butler, PhD, Principal Investigator — University of California, Davis